CLINICAL TRIAL: NCT06785753
Title: Effectiveness of Intracanal Cryotherapy on Post Operative Pain After Root Canal Therapy in Patients with Symptomatic Apical Periodontitis
Brief Title: Effectiveness of Cryotherapy on Endodontic Pain
Acronym: Cy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Hira Amjad, Dr. Hira Amjad , Principal investigator and Resident Operative Dentistry and Endodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cryotherapy
Record Dates: First submitted 2023-06-10; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- normal saline group (Experimental): In control group , canals will be irrigated with 5ml of normal saline at room temperature
  Interventions: Drug: Irrigation Solution
- cryotherapy (cold saline group) (Experimental): in cold saline group , canals will be irrigated with 5 ml of cold saline at a temperature of 2.5° C
  Interventions: Drug: Irrigation Solution

INTERVENTIONS:
Drug: Irrigation Solution — normal saline will be used as irrigation solution
  Other Names: normal saline irrigant

SUMMARY:
This is a randomized , prospective , control trial to assess the effectiveness of intracanal cryotherapy on post operative pain after root canal treatment in patients with symptomatic apical periodontitis

DETAILED DESCRIPTION:
Diagnostic procedures to include patients history taking , clinical and radiographic with all findings being recorded in patients .

patients diagnosed with symptomatic irreversible pulpitis with symptomatic apical periodontitis.

patients will be asked to rate their pre treatment pain on visual analogue scale from 0-10

patients with pain score <8 will be considered

Anesthesia and isolation : after administration of local anesthesia , rubber dam application will be done

Acess cavity : acess will be gained with round bur using air turbune handpiece with copious water cooling

Working length : a size 10k file will be inserted into the canal to determine the working length with the help of radiograph

Cleaning and shaping : Extirpation of pulp will be done followed by canal preparation with manual and endodontic motor using naocl and EDTA .

final irrigation will be performed using 17% EDTA and 5.25% NaOCl

Patients will be divided into 2 group in control group : final irrigation will be done using 5ml of saline at room temperature in cold group : final irrigation will be done using 5ml of cold saline at 2.5°C

the solution will be stored in the refrigerator until use irrigation will be performed for 5 min in both groups using 27 G beveled needle tip inserted 2mm short of WL.

Obturation ; In both groups , canals will be dried with paper points and obturated using gutta percha cones with zinc oxide eugenol sealer

Restoration : acces cavity will be restroed with direct composite restoration or high viscosity glass ionomer cement

each patient will be given instruction to acess the post operative pain .

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic irreversible pulpitis and symptomatic apical periodontitis
* maxillary or mandibular single rooted teeth
* systemically healthy patients
* patients having pain score < 8

Exclusion Criteria:

* patients on preoperative analgesics or antibiotics within past 12 hours
* teeth with calcified canals and previously treated teeth
* tooth with immature apices or resorption
* patients allergic to local anesthesia
* pregnant or lactating mothers
* patients who are immunocompromised .

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-05-07 (Estimated); Study Completion 2025-05-08 (Estimated)

PRIMARY OUTCOMES:
post operative pain after root canal treatment | 1 week
  post operative pain will be assessed using visual analogue scale ( VAS) from 0-10 each patient will be given instruction to access the post operative pain . it will be carried out using a questionnaire.
  VAS 0-1 = No pain 2-3 = mild pain 4-6 = moderate pain 7-10 = severe pain pain recording will be done at 6 hrs , 24 hrs, 48hrs and 72 hrs. ( participants to be contacted by investigator at each point to check on them and remind them to record their pain ). The given questionnaire shall be collected when the participant comes for final restoration after 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Hira Amjad, BDS, Principal Investigator — Armed Forces Institude Of Dentistry
Locations (1):
- Armed Forces Institute of Dentistry, Rawalpindi, Punjab Province, Pakistan